CLINICAL TRIAL: NCT01023867
Title: Comparative Assessment of Clinical Efficacy of Donepezil Between the Patients With Alzheimer's Disease and Mixed Dementia
Brief Title: Clinical Trial of Donepezil Between the Patients With Alzheimer's Disease and Mixed Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Eisai Korea Inc. (Industry)
Responsible Party: Principal Investigator, Doh Kwan Kim, Professor, Samsung Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007-03-039
Record Dates: First submitted 2009-11-30; First posted 2009-12-02 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2016-01

CONDITIONS: Alzheimer's Disease; Dementia
Keywords: Alzheimer's disease; Mixed Dementia; Donepezil; Efficacy; Adverse Event
MeSH Terms: conditions — Alzheimer Disease; Dementia; Mixed Dementias | interventions — Donepezil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alzheimer's disease group (Experimental): Patients with Alzheimer's disease treated donepezil
  Interventions: Drug: donepezil
- Mixed Dementia group (Experimental): Patients with Mixed Dementia treated donepezil
  Interventions: Drug: donepezil

INTERVENTIONS:
Drug: donepezil — from 5mg to 10mg, once a day, 12 months
  Other Names: donepezil-aricept

SUMMARY:
To compare the clinical efficacy of donepezil between patients with Alzheimer's disease and Mixed Dementia.

DETAILED DESCRIPTION:
The purposes of this study are:

1. to compare the clinical efficacy of donepezil between patients with Alzheimer's disease and Mixed Dementia
2. to help to clinicians in choosing the best treatment for patients with mixed dementia

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of probable AD and Mixed Dementia according to the criteria of the NINCDS-ADRDA
2. Korean version Mini-Mental State Examination scores between 10 and 26
3. History of cognitive decline that had been gradual in onset and progressive over at least 6 months
4. A caregiver who could assist the patient with medication, attend the assessment and provide information about the patient.

Exclusion Criteria:

1. they had evidence of any neurodegenerative diseases other than AD (i.e. Parkinson's disease, Huntington's disease)
2. Psychiatric disorder or severe behavioral disturbances that required psychotropic medications
3. Cerebral injuries induced by trauma, hypoxia, and/or ischemia
4. Clinically active cerebrovascular disease; History of seizure disorder
5. Other physical conditions that required acute treatment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2007-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale-Cognitive, Korean version (ADAS-Cog-K) | 13 weeks, 26 weeks, 39 weeks, 52 weeks

SECONDARY OUTCOMES:
Seoul Activities of Daily Living (S-ADL) | 13 weeks, 26 weeks, 39 weeks, 52 weeks
Seoul-Instrumental Activities of Daily Living (S-IADL) | 13 weeks, 26 weeks, 39 weeks, 52 weeks
Korean Neuropsychiatric Inventory (K-NPI) | 13 weeks, 26 weeks, 39 weeks, 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Doh Kwan Kim, PhD, M.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea